CLINICAL TRIAL: NCT05910320
Title: Evaluation of an Investigational Wearable Vital Signs Monitoring Device in Healthy Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed at site. Investigator no longer at site.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00361015
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable Vital Signs Monitoring Device (Experimental)
  Interventions: Device: Wearable Vital Signs Monitoring Device

INTERVENTIONS:
Device: Wearable Vital Signs Monitoring Device — The prototype will be used to non-invasively measure vital signs. This prototype (preliminary version) is composed of a sensor module, a rechargeable battery, and electrodes. The device is housed in a waterproof, silicone casing.

SUMMARY:
The primary objective of this study is to evaluate the feasibility of the use of an investigational wearable vital sign monitoring device in infants.

DETAILED DESCRIPTION:
Vital sign monitoring of infants outside of a traditional healthcare setting has already been shown to significantly decrease mortality for children with single ventricle congenital heart disease (1V CHD), a fragile group of patients with congenital heart disease (CHD). Therefore, there is a critical need to develop an accurate, at-home vital sign monitoring system for infants to expand the benefits of remote monitoring to further patient populations. The investigators believe that allowing for continuous monitoring at a clinical standard with interpretations and alerts built into the technology will result in an even greater decline in mortality for infants with 1V CHD, improved clinical outcomes for all infants with CHD, and increased well-being for healthy infants.

To achieve this goal, the investigators are developing a health monitoring system that collects numerical data and physiological waveforms describing heart rate (HR), respiratory rate (RR), pulse oximetry (SpO2), regional oxygen saturation, temperature, and infant motion.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to either the newborn nursery, pediatric cardiac intensive care unit (PCICU), or pediatric care unit (PCU)
* Parent provided written informed consent

Exclusion Criteria:

* Foster or ward of the state

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Signal morphology of wearable monitoring device | From device placement to removal, up to 1 hour
  Feasibility of a wearable monitoring device as determined by signal morphology of wearable monitoring device
Signal-to-noise ratio of wearable monitoring device | From device placement to removal, up to 1 hour
  Feasibility of a wearable monitoring device as determined by signal-to-noise ratio
Signal-to-noise ratio of reusable electrodes | From electrode placement to removal, up to 15 minutes
  Feasibility of reusable electrodes as determined by the signal-to-noise ratio
Percent error of wearable monitoring device compared to clinical bedside monitors | From device placement to removal, up to 1 hour
  Feasibility of a wearable monitoring device as determined by percent error compared to clinical bedside monitors

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Gottlieb Sen, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States